CLINICAL TRIAL: NCT01748877
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Tolerability, and Safety of NXN-462 in Patients With Post-Herpetic Neuralgia (PHN)
Brief Title: Efficacy, Tolerability, and Safety of NXN-462 in Patients With Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurAxon Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NXN-462-201
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Post Herpetic Neuralgia
Keywords: shingles,; neuropathic pain; post herpetic neuralgia; sleep
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NXN-462 (Experimental): capsule, 200 mg, bi.d. 28-days
  Interventions: Drug: NXN-462
- Placebo (Placebo Comparator): capsule, b.i.d. 28-days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NXN-462 — Study drug is to be self-administered twice each day by the patient. Each day the first dose of study drug should be taken preferably one hour prior to, OR one hour after the first meal (breakfast) of the day. The second and final dose each day should be taken with a glass of water at least one hour after the last meal immediately before retiring to sleep.
  Other Names: NXN-462 dihydrochloride
  Arms: NXN-462
Drug: Placebo — Study drug is to be self-administered twice each day by the patient. Each day the first dose of study drug should be taken preferably one hour prior to, OR one hour after the first meal (breakfast) of the day. The second and final dose each day should be taken with a glass of water at least one hour after the last meal immediately before retiring to sleep.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether NXN-462, a selective nNOS inhibitor, is effective in reducing pain levels in patients with post-herpetic neuralgia.

DETAILED DESCRIPTION:
NXN-462 is designed to target the nitric oxide synthase system (NOS), specifically the neuronal NOS (nNOS) isoform. By design, NXN-462 is a potent inhibitor of nNOS with good affinity, and has little or no affinity for a range of G protein-coupled receptors, ion channels, and enzymes. NXN-462 is being developed as an oral therapy for the treatment of neuropathic pain syndromes, including PHN. This drug design strategy provides a new therapeutic paradigm for the treatment of chronic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male, or a non-pregnant, non-lactating female 18 years or older
* Have voluntarily provided written informed consent
* able to speak, read, write, and understand English
* clinical diagnosis of PHN for a minimum of 6 months
* pain intensity score of ≥3 on a 0-10 Numerical Rating Scale (NRS) at the Screening Visit
* generally in good health (other than PHN) at Screening

Exclusion Criteria:

* Are pregnant and/or lactating
* Diagnosis of any chronic pain syndrome that would interfere with the assessment of PHN
* evidence of multiple causes of neuropathic pain,e.g.lumbar radiculopathy in the lumbosacral area
* Have had neuroablation or neurosurgical intervention for PHN
* Have been taking opioid analgesics for >5 days/week
* Have received nerve block or intrathecal analgesia within 6 weeks of the study
* History of significant gastrointestinal disease, liver disease, renal disease, endocrine disease, or cardiovascular disease
* clinically significant abnormal clinical laboratory test results or vital signs
* Are immunocompromised or immunosuppressed for any reason
* History of alcohol or other substance abuse (not including nicotine or tobacco) within 5 years
* Significant psychiatric disorder which requires drug treatment (except depression or anxiety treated with Selective Serotonin Re-uptake Inhibitors)
* Have received an investigational drug or have used an investigational device within 30 days of Screening.
* Have previously been randomized to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the last week of treatment in daily pain scores | 4 weeks
  Change from baseline to the last week of treatment in daily (24-hour recall) pain scores comparing NXN-462 with placebo

SECONDARY OUTCOMES:
average weekly change in pain score from baseline to the end of the Treatment Period | four weeks
Analysis of percent change from baseline in daily pain score | four weeks
percentage of responders | four weeks
  subjects with a ≥30% and ≥50% reduction in pain score from baseline to the last week of treatment
Percentage of subjects with moderate or much improvement at the end of the Treatment Period, according to Patient Global Impression of Change | four weeks
Change from baseline to the end of the Treatment Period in Pain Quality Assessment Scale score | four weeks
Rescue medication consumption | four weeks
Adverse events (AEs), vital signs, and clinical laboratory tests | six weeks
Change from baseline to the end of the Treatment Period in Modified Brief Pain Inventory Short Form score, pain interference subscale | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lategan, D.Phil., Study Director — NeurAxon Inc.
Locations (25):
- United States (22):
  - Premier Research, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Northern California Research, Sacramento, California
  - Neurological Research Institute, Santa Monica, California
  - Meridien Research, Brooksville, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Compass Research LLC, Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Integrated Clinical Trial Services, West Des Moines, Iowa
  - IRC Clinics, Towson, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Michigan Head-Pain and Neurological Institute, Ann Arbor, Michigan
  - Albuquerque Clinical Trials, Inc, Albuquerque, New Mexico
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Pain Specialist of Charleston, P.A., Mt. Pleasant, South Carolina
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Trinity Clinical Research, Tullahoma, Tennessee
  - ClinRx Research LLC, Plano, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Canada (3):
  - Manna Research Vancouver, Vancouver, British Columbia
  - Manna Research, Inc., Toronto, Ontario
  - Kells Medical Research Group - Manna Research, Pointe-Claire, Quebec